CLINICAL TRIAL: NCT00877019
Title: Time Dependent Professional Toothbrushing Study Comparing Sonicare With Manual Toothbrushes
Brief Title: Time Dependent Professional Toothbrushing Study
Acronym: timebrush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: PD Dr. M. PElka, Dental Clinic 1 - Operative Dentistry and Periodontology, University of Erlangen-Nürnberg
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Toothbrushing
Keywords: sonic brushes; time effectiveness; brush head design; ADA-toothbrush; professional brushing; time dependence; efficacy; toothbrush

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Sonicare elite medium brush head
Device: Sonicare elite mini brushhead
Device: GABA Elmex sensitive extra soft toothbrush
Device: ADA reference toothbrush

SUMMARY:
Aim:

The study was designed to test the time dependent efficacy in plaque removal of four toothbrushes: one electric toothbrush, the Philips Sonicare Elite with long (A) and short (B) brushing head and two manual brushes, the Gaba Sensitve (C), and the ADA reference brush (D) and.

Materials and Methods:

The study was a single-blind, randomized clinical timer study consisting of four identical experiments testing each brush in one quadrant. The distribution of the quadrants and brushes was randomized so that always all brushes were used within one participant. The teeth were brushed by a dental hygienist for 10, 20, 30, 45, 60 und 90 seconds per quadrant. No toothpaste was used throughout this study. The plaque assessment (Tureskey modified QHI) was done after each time interval blinded on six sites per tooth by a separate investigator. Ninety subjects participated in the study and received a professional prophylaxis prior to the experiment. They were requested to refrain from brushing their teeth for 48 hours prior to the experiment.

ELIGIBILITY:
Inclusion Criteria:

* at least 24 evaluable teeth in the mouth

Exclusion Criteria:

* systemic disease
* regular drugs or actual antibiotics
* orthodontic banding or retention wires
* oral lesions or sites with a probing pocket depth X5 mm

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)